CLINICAL TRIAL: NCT07229885
Title: Comparison of Early Versus Late Trophic Feeding in Preterm Very Low Birth Weight Neonates at a Tertiary Care Hospital
Brief Title: Comparison of Early Versus Late Trophic Feeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RESnTEC, Institute of Research (Other)
Responsible Party: Principal Investigator, Muhammad Aamir Latif, Research Consultant, RESnTEC, Institute of Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dr-Nadeem-Nishter
Record Dates: First submitted 2025-09-30; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Very Low Birth Weight Infant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early trophic feeding group (Experimental): Infants will receive trophic (enteral) feeding within the first 48 hours after birth.
  Interventions: Dietary Supplement: Early trophic feeding
- Late trophic feeding group (Experimental): Infants will receive trophic (enteral) feeding after 72 hours after birth.
  Interventions: Dietary Supplement: Late trophic feeding

INTERVENTIONS:
Dietary Supplement: Early trophic feeding — Infants will receive trophic (enteral) feeding within the first 48 hours after birth.
  Arms: Early trophic feeding group
Dietary Supplement: Late trophic feeding — Infants will receive trophic (enteral) feeding within the first 72 hours after birth.
  Arms: Late trophic feeding group

SUMMARY:
Local data on the neonatal outcomes in early versus late trophic feeding in preterm very low birth weight neonates in terms of mean hospital stay is scarce. Therefore, the current study was planned with the objective of comparing the neonatal outcomes in early versus late trophic feeding in preterm very low birth weight neonates in terms of mean hospital stay.

DETAILED DESCRIPTION:
Since preterm, very low birth weight births are common in society, an effective treatment modality is needed at the moment. Evaluating the length of hospital stay and occurrence of necrotizing enterocolitis in preterm very low birth weight neonates with respect to two approaches of trophic feeding in local settings will provide an insight into a better implementation of preventive strategies, resulting in reducing the hospital stays and the incidence of necrotizing enterocolitis, and hence reducing the burden on the already meager resources.

ELIGIBILITY:
Inclusion Criteria:

* Any gender
* Neonates aged 1-30 days
* Preterm very low birth weight neonates

Exclusion Criteria:

* Neonates transferred from other hospital and already started on antibiotics.
* Neonates with congenital anomalies, hypoxic ischemic encephalopathy, central nervous system (CNS) impairment, neonatal sepsis, urinary tract infection, or one of twins or higher order multiples (on history and medical record).
* Non-consenting parents.

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Incidence of necrotizing enterocolitis | Up to 30 days
  Confirmation of the occurrence of necrotizing enterocolitis based on modified Bell's diagnostic criteria

SECONDARY OUTCOMES:
Hospital stay | through study completion, an average of 1 month
  Total days from admission till final outcome (discharge/death due to any case).

CONTACTS AND LOCATIONS:
Overall Officials: Nadeem Akram, Principal Investigator — Nishter Hospital Multan, Pakistan; Sulaiman Ali, FCPS, Study Director — Nishter Hospital Multan, Pakistan
Locations (1):
- Nishtar Hospital, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
Data can be shared on a reasonable request.